CLINICAL TRIAL: NCT00244413
Title: Nondystrophic Myotonias: Genotype-phenotype Correlation and Longitudinal Study
Brief Title: Characteristics of Nondystrophic Myotonias
Status: Completed | Type: Observational
Sponsor: Richard Barohn, MD (Other)
Collaborators: Office of Rare Diseases (ORD) (NIH); Rare Diseases Clinical Research Network (Network)
Responsible Party: Sponsor-Investigator, Richard Barohn, MD, Gertrude and Dewey Zeigler Professor of Neurology and Chair, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Other Study IDs: 10263
Record Dates: First submitted 2005-10-24; First posted 2005-10-26 (Estimated); Last update posted 2013-03-06 (Estimated); Status verified 2013-03

CONDITIONS: Nondystrophic Myotonias; Myotonia Congenita; Myotonic Disorders
Keywords: Myotonia; Paramyotonia Congenita; Thomsen's Disease
MeSH Terms: conditions — Myotonia Congenita; Myotonic Disorders; Myotonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples

SUMMARY:
Nondystrophic myotonias (NDM) are muscle disorders caused by genetic abnormalities in certain muscle cell membrane proteins. Individuals with NDM experience limited muscle relaxation, which causes pain, weakness, and impaired physical activity. The purpose of this study is to better characterize the clinical features and symptoms of NDM.

DETAILED DESCRIPTION:
Nondystrophic myotonias are muscle disorders caused by abnormal muscle cell membrane proteins that affect the control of muscle fiber contraction. These disorders are extremely rare, and little is known about how to best treat the various subtypes of NDM. The purpose of this study is to characterize the clinical features and symptoms of NDM as well as to pair this data with specific NDM subtypes. In turn, this may lead to the development of improved treatments. The study will also establish clinical endpoints for use in future studies.

This multi-center observational study will involve both a cross-sectional data analysis and a prospective longitudinal analysis. Participants will initially attend a one-day outpatient study visit. Various baseline measurements will be collected, including demographics, medical history, and quality of life measures. Blood samples will be taken to evaluate laboratory values and genetic factors. Participants will undergo manual muscle testing (MMT), clinical myotonia assessments, and functional movement assessments. Routine nerve conduction studies and electromyography (EMG) will also be performed in order to test for the presence of myotonia in specific muscles. Annual follow-up evaluations will occur 1 and 2 years following the first study visit.

ELIGIBILITY:
Inclusion Criteria:

* Clinical symptoms or signs suggestive of myotonia
* Presence of myotonic potentials on electromyography (EMG)
* Persistence of symptoms and signs after discontinuation of medications that produce myotonia; such medications include fibric acid derivatives, hydroxymethylglutaryl CoA reductase inhibitors, chloroquine, and colchicine
* Absence of features suggestive of myotonic dystrophy, including ptosis, temporal wasting, mandibular weakness, cataracts occurring before age 50, and evidence of multisystem defects (cardiac conduction defects, hypogonadism)

Exclusion Criteria:

* Any other neurologic condition that might affect the assessment of the study measurements

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with nondystrophic myotonia
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2006-02; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Examine the frequency applicable events related to Nondystrophic Myotonia | Baseline - 3 yrs
  We will measure by an interactive voice response to measure stiffness, pain, weakness, and fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Barohn, MD, Principal Investigator — University of Kansas Medical Center
Locations (6):
- United States (4):
  - University of Kansas Medical Center, Department of Neurology, Kansas City, Kansas
  - Brigham & Women's Hospital, Department of Neurology, Boston, Massachusetts
  - University of Rochester School of Medicine and Dentistry, Department of Neurology, Rochester, New York
  - University of Texas Southwestern Medical Center, Dallas, Texas
- London Health Sciences Centre, University Hospital, London, Ontario, Canada
- Center for Neuromuscular Disease, Institute of Neurology and National Hospital for Neurology, London, United Kingdom

REFERENCES:
- [Background] Torbergsen T, Hodnebo A, Brautaset NJ, Loseth S, Stalberg E. A rare form of painful nondystrophic myotonia. Clin Neurophysiol. 2003 Dec;114(12):2347-54. doi: 10.1016/s1388-2457(03)00275-x. PMID 14652094
- [Background] Renner DR, Ptacek LJ. Periodic paralyses and nondystrophic myotonias. Adv Neurol. 2002;88:235-52. No abstract available. PMID 11908229
- [Background] Cannon SC. Spectrum of sodium channel disturbances in the nondystrophic myotonias and periodic paralyses. Kidney Int. 2000 Mar;57(3):772-9. doi: 10.1046/j.1523-1755.2000.00914.x. PMID 10720928
- [Background] Cannon SC. From mutation to myotonia in sodium channel disorders. Neuromuscul Disord. 1997 Jun;7(4):241-9. doi: 10.1016/s0960-8966(97)00430-6. PMID 9196906
- [Background] Moxley RT 3rd. The myotonias: their diagnosis and treatment. Compr Ther. 1996 Jan;22(1):8-21. No abstract available. PMID 8654027
- [Background] Brown RH Jr. Ion channel mutations in periodic paralysis and related myotonic diseases. Ann N Y Acad Sci. 1993 Dec 20;707:305-16. doi: 10.1111/j.1749-6632.1993.tb38061.x. No abstract available. PMID 9137561